CLINICAL TRIAL: NCT04835545
Title: Work of Breathing Under Extreme Hypercapnia Induced by Ventilation Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DP-2021-Nemec
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Accident Caused by Snow Avalanche
Keywords: snow; avalanche; hypercapnia; work of breathing
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wet Perlite, 2L air pocket (Experimental): Breathing in the simulated avalanche snow. Breathing into model of wet perlite with 2L air pocket
  Interventions: Other: extreme hypercapnia induced by ventilation insufficiency
- Wet Perlite 2L air pocket with resistance compensation (Experimental): Breathing in the simulated avalanche snow. Breathing into model of wet perlite 2L air pocket with resistance compensation
  Interventions: Other: extreme hypercapnia induced by ventilation insufficiency
- Wet Perlite, no air pocket (Experimental): Breathing in the simulated avalanche snow. Breathing into model of wet perlite with no air pocket
  Interventions: Other: extreme hypercapnia induced by ventilation insufficiency

INTERVENTIONS:
Other: extreme hypercapnia induced by ventilation insufficiency — extreme hypercapnia

SUMMARY:
The aim of the study is to investigate Work of Breathing of a person in simulated avalanche snow and consequent use of the measured data for judging which one of three simulated scenarios are alike while increasing hypercapnia in the simulated avalanche snow.

DETAILED DESCRIPTION:
The study is a part of a university diploma thesis aimed at studying physiological conditions and development of breathing parameters of a person breathing in the simulated avalanche snow. The Investigator is measuring Work of Breathing in three scenarios: a) 2L air pocket, b) 2L air pocket with resistance compensation and c) no air pocket. The investigator hypothesize that the Work of Breathing during compensation of air pocket will be alike with no air pocket scenario, thus proving significance of the resistance reduction for survival. The aim of the study is to investigate the effect of Work of Breathing on gas exchange in subjects breathing into the simulated avalanche snow scenarios.

ELIGIBILITY:
Inclusion Criteria:

* healthy and fit volunteers, classified as The American Society of Anesthesiologists class I
* without a smoking history

Exclusion Criteria:

* Tiffeneau Index less than 0.70
* any cardiovascular or respiratory condition

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The length of breathing | Continuously within up to 7 minute interval from the beginning of the breathing experiment
  Time to termination of the breathing experiment due to the decision of the tested subject, or determined by high end-tidal carbon dioxide value or by the order by the clinician assessing the health status of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubík, PhD, Study Director — Czech Technical University in Prague, FBMI
Locations (1):
- Czech Technical University, Faculty of Biomedical Engineering, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roubik K, Sieger L, Sykora K. Work of Breathing into Snow in the Presence versus Absence of an Artificial Air Pocket Affects Hypoxia and Hypercapnia of a Victim Covered with Avalanche Snow: A Randomized Double Blind Crossover Study. PLoS One. 2015 Dec 14;10(12):e0144332. doi: 10.1371/journal.pone.0144332. eCollection 2015. PMID 26666523